CLINICAL TRIAL: NCT04215367
Title: Effect of Dietary Intervention With High-Oleocanthal and Oleacin Extra Virgin Olive Oil in Patients With Chronic Lymphocytic Leukemia a Pilot Study
Brief Title: Dietary Intervention With High Phenolic EVOO in CLL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Peloponnese (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Harokopio University (Other)
Responsible Party: Principal Investigator, Andrea Paola Rojas Gil, Assistant Professor, University of Peloponnese
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 44917/13-12-2018
Record Dates: First submitted 2019-12-07; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: CLL; oleocanthal; Extra Virgin Olive Oil (EVOO); phenols; apoptosis
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: Twenty one patients with Chronic lymphocytic leukemia (CLL) from the hematologic clinic of the General hospital of LaKonia (Greece), were enrolled to participate in the dietary intervention. CLL diagnosis was confirmed by standard criteria. Patients were untreated, in Rai stage 0 to II, did not met criteria to initiate chemotherapy and had no neoplasmatic comorbidity. Subjects were randomly selected from the Hematology Department of the General Hospital of Lakonia. Exclusion criteria were neoplastic comorbidities or severe metabolic diseases. Only one group participates in this study, which performed dietary intervention consuming EVOO rich in oleocanthal and oleacin. Clinical and molecular markers were registered 6 months before the intervention and 6 months during the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High phenolic EVOO intake (Experimental): Patients with CLL consumed before their meals, 40 ml/day of EVOO rich in oleocanthal and oleacin for 6 months,
  Interventions: Dietary Supplement: High phenolic EVOO intake
- No High phenolic EVOO intake (Experimental): Patient's history were recorded for third and sixth month before dietary the intervention, taking into consideration that the patients did'nt consume high phenolic EVOO.
  Interventions: Dietary Supplement: No High phenolic EVOO intake

INTERVENTIONS:
Dietary Supplement: High phenolic EVOO intake — During the pilot dietary intervention patients with CLL consumed before their meals, 40 ml/day high phenolic EVOO for 6 months
  Arms: High phenolic EVOO intake
Dietary Supplement: No High phenolic EVOO intake — Medical record of each patient's was followed during 6 month before dietary the intervention
  Arms: No High phenolic EVOO intake

SUMMARY:
Daily intake of extra virgin olive oil (EVOO), which is the major component of the Mediterranean diet and also a source of monounsaturated fat, may be partly responsible for the increased life expectancy of the Mediterranean people. A high dietary intake of EVOO is correlated with lower incidence of cancer, cardiovascular disease, metabolic diseases, Alzheimer's disease and osteoporosis Oleocanthal, a phenolic derivative of extra virgin olive oil, has important health promoting anti-cancerous properties, since it can inhibit the growth and promote the apoptosis of several cancer cells.

The purpose of the present study was to investigate the effect of dietary intake of olive oil rich in oleocanthal on hematological, metabolical, cell progression markers and disease progression in patients with Chronic Lymphocytic Leukemia. The aim is also to study the possible association of apoptosis in the mechanism of action of virgin olive oil phenols in a patient with CLL in order to find the possible mechanism of the cellular action of oleocanthal in neoplasia.

After the screening of >300 EVOO samples the investigators selected an EVOO with high oleocanthal and oleacin concentration of 416 and 284 mg/Kg respectively (EVOO OC/OL). Pilot dietary intervention was made in a group of 21 patients with chronic lymphocytic leukemia (CLL) who did not follow any treatment. EVOO was administered 40 ml/day for six months. Biochemical, hematological and molecular markers were studied six month before the intervention and six month during the intervention

DETAILED DESCRIPTION:
Extra virgin olive oil (EVOO) is the major component of the Mediterranean diet. More than 200 different chemical compounds have been detected in olive oil, including fatty acids, sterols, carotenoids, terpenoids, flavonoids, tocopherols and olive polyphenols. Virgin olive oil contains a variety of important phenolic components, mainly corresponding to the compounds tyrosol, hydroxytyrosol, oleocanthal (OC) ,oleacin (OL) ,ligstroside and oleuropein aglycones .Among these olive phenols, oleocanthal , a dialdehydic form of dicarboxymethyl ligstroside aglycone which has been isolated from EVOO, presents a wide range of biological effects including antioxidant, anti-inflammatory, anticancer, neuroprotective and antidiabetic activities and for this reason has attracted more scientific attention.

Chronic Lymphocytic Leukemia (CLL), the most commonly diagnosed adult leukemia in Western countries, is responsible for about 1 in 4 cases of all leukemias. It is characterized by the accumulation of monoclonal B-cells in bone marrow, peripheral blood, lymphatic tissues and spleen, while it is often asymptomatic and slow in its development. Patients with CLL do not always require immediate therapy. However, patients who appear symptoms have an approximate median survival range from 18 months to 6 years depending on the clinical stage. Criteria for the diagnosis of CLL are monoclonal B lymphocytes ≥5000 lymphocytes/ml in the peripheral blood for at least 3 months, prolymphocytes ≤55%, co-expression of claster of diferentiation (CD)5 and B-cell surface antigens CD 19, CD 20, and CD 23, low levels of CD 20, CD 79b and low expression of surface immunoglobulins (sIg), and kappa or lambda light chain restriction. The standard clinical procedures to estimate prognosis are the clinical staging systems developed by Rai et al and Binet et al.

The level of apoptosis in hematopoiesis may provide information about the mechanism which is responsible for the regulation of progenitor's and stem cell's proliferation. The dysfunction of apoptosis has found to be associated with leukemia. An increase in the expression of Apo-1/fas (CD 95) apoptotic marker in myeloid progenitor cells in CLL patients and a corresponding decrease in the apoptotic B-cell lymphoma 2 (BCL-2) inhibitor has been described. Recent studies showed also that the increase in CLL patients' lymphocytes may be due to the disturbed balance between the proliferation and apoptosis of CLL cells while the changes in apoptosis-related protein expression are recognized during all the stages of Binet in CLL. The p38 levels are reduced (resistance to apoptosis) and Induced myeloid leukemia cell differentiation protein (Mcl-1) and Survivin levels are elevated, so as to enhance the survival of B lymphocytes.

Survivin is a protein inhibitor of apoptosis which inhibits caspases and blocks cell death. It is highly expressed in most cancers, including hematological, and is associated with a poor clinical outcome. The apoptotic marker CD 95 (Apo-1/fas) and its ligand, CD 95 is a death receptor ligand that mediates apoptosis induction in order to maintain immune homeostasis and has the capacity to mediate apoptosis induction in cancer cells, generating an 18-kilodalton fragment termed caspase-cleaved cytokeratin-18 (cCK-18).

Oleocanthal has been shown to induce cytotoxicity and apoptosis in vitro in human acute promyelocytic leukemia and in myeloma cells. It may also cause primary necrosis and cellular apoptosis by inducing lysosomal membrane permeability in different cancer cell lines.

The aim of this study taking into account the strong apoptotic properties of oleocanthal in vitro, was to investigate its ability, under real clinical settings, to affect the hematological and biochemical profile; also the cellular apoptotic markers Survivin, cCK18- (caspase activity marker) and Apo1fas/CD 95 in CLL patients after taking into consideration the progression of their disease. For this reason was conducted a dietary intervention study comparing the antineoplastic effects of an oleocanthal-rich EVOO in CLL patients.

Material and Methods

In the current study, a screening of 300 commercial samples (selected among a database of >3000 samples), obtained from olives (Olea europaea L.) harvested in 2017-2018 season, was performed by the Quantitative NMR spectroscopy (qNMR) method in order to identify oils which could fulfill the following criteria: The extravirgin oil would have high oleocanthal and oleacin content (D1 index) and low or even no content in other secoiridoid conjugated phenolics (3-8) or free tyrosol and hydroxytyrosol Specifically Oil rich in Oleocanthal was obtained from Monovarietal oil of Lianolia Kerkyras variety provided by "The Governor" Company from Agios Matthaios, Corfu, Greece. This oil contained: Oleocanthal 416±7 mg/Kg, oleacin 284±10 mg/Kg, Tyrosol < 10 mg/Kg, Hydroxytyrosol < 10 mg/Kg (D1 = 700 mg/Kg). It should be mentioned that apart the qNMR analysis, the hydroxytyrosol and tyrosol content was also measured by the standard IOC method for measurement of olive oil biophenols. Selected EVOO immediately after their analysis and until the beginning of the study period were stored at 4 celsious degree in order to minimize possible alterations in chemical composition.

Subjects Twenty one patients from the hematologic clinic of the General hospital of Lakonia (Greece), were enrolled to participate in the dietary intervention. CLL diagnosis was confirmed by standard criteria. Patients were untreated, in Rai stage 0 to II.

Dietary Intervention At the begin of the pilot study medical exams of each patient's history were recorded for third and sixth month before dietary the intervention. The clinical record before the dietary intervention concerns the hematological profile, biochemical exams including, lipidemic profile, fasting glucose, Liver and kidney function markers, as well as data concerning blood marrow biopsy, neoplastic markers and immunophenotype. Drug treatment or comorbidities were also recorded.

At the begin of the pilot dietary intervention a group of 21 patients with CLL consumed before their meals, 40 ml/day of EVOO rich in olecanthal and oleacin (OC/OL) for 6 months, in order to explore the effect of the dietary consumption of the A-EVOO on the studied hematological, biochemical and molecular markers. The amount of the consumed EVOO OC/OL was chosen according to a previous study. (15) Patients were advised to continue their regular diet; their adherence to the study protocol was assessed by two 24-h telephone recalls every two weeks.

Peripheral blood samples from the 21 patients with CLL were gathered at the begin, after 3 months and after 6 months from the begin of the dietary intervention. Whole blood count and complete biochemical tests were performed for fasting glucose, blood lipid profile, and markers of liver and kidney function. Serum analyses were conducted using the same procedure and at the same lab with the use of a biochemical analyzer (Olympus AU-600, Olympus, Tokyo, Japan).

A commercially available enzyme-linked immunosorbent assay (ELISA) was used according to the instructions of the supplier to assay the apoptotic markers M30 Apoptosense-cCK18 (VLVbio Hästholmsvägen, Sweden), Apo-1/Fas/CD 95 (Novus Biologicals, Colorado USA) and the antiapoptotic marker Survivin (OriGene Technologies, Inc USA) into plasma samples of all the patients at all the studied time points.

Statistical analysis was performed using SPSS v.24 (SPSS Inc., Chicago, IL. USA) and the significance level was set at 0.05. Initially a descriptive analysis of the sample was performed in terms of age, sex, clinical, biochemical and molecular markers. The markers were found to be skewed at p < 0.05 significance level when checked by using the Kolmogorov-Smirnov test. Therefore non-parametric Mann-Whitney U test were used to find out the differences between the intervention and the control group.

The differences between the time intervals of the intervention was assessed with Friedman non-parametric test followed by Dunn's test for multiple comparison Finally, the correlations of the molecular markers with the clinical parameters included in the study and were checked with Spearman Rho.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Chronic lymphocytic leukemia (CLL)
* Untreated CLL patients having Rai stage 0 to II
* Must be able to consume high phenolic EVOO according to the instructions

Exclusion Criteria:

* Neoplasic comorbidities and received any chemotherapy,
* Severe metabolic disease such us insulin dependent diabetes or severe kidney disease

Ages: 54 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Effect of the dietary intake of high phenolic EVOO on hematologic profile | 1 year
  The effect of the dietary intake of high phenolic EVOO on hematologic profile was investigated comparing the complete blood count before (6 and 3 months) at the starting point of the dietary intervention and during (3 and 6 months) the dietary intervention in order to evaluate possible sustained hematologic improvement according to Rai et al criteria. Whole cell blood account was evaluated by hematological analyzer.
Effect of the dietary intake of high phenolic EVOO on apoptotic markers | 6 month
  The effect of the dietary intake of high phenolic EVOO on apoptotic markers was investigated comparing the protein expression level on serum of the participants by ELISA. The apoptotic proteins Apo-1/Fas CD 95 (pg/ml) and CCK18 (U/L) and the antiapoptotic protein Survivin (pg/ml) were studied. The mentioned markers were evaluated at the starting point of the intervention, at 3 and 6 months during the dietary intervention with high phenolic EVOO in order to evaluate the in vivo the effect of high phenolic EVOO on protein expression of the studied apoptotic markers in CLL.

SECONDARY OUTCOMES:
Effect of the dietary intake of high phenolic EVOO on fasting glucose and correlation with the clinical outcome of the patients with CLL | 1 year
  The effect of the dietary intake of high phenolic EVOO on fasting glucose (mg/dL), was investigated comparing the fasting glucose before the intervention (6 and 3 months) at the starting point of the intervention, at 3 and 6 months during the dietary intervention with high phenolic EVOO. The correlation of the changes on the fasting glucose during the survey with the hematological outcome of the patient with CLL was also investigated.
Effect of the dietary intake of high phenolic EVOO on lipidemic profile and correlation with the clinical outcome of the patients with CLL | 1 year
  The effect of the dietary intake of high phenolic EVOO on lipidemic profile (cholesterol (mg/dl), Low density lipoprotein (LDL- mg/dl), Hight density lipoprotein (HDL mg/dl), tryglicerides (mg/dl) was investigated comparing the lipidemic profile before the intervention (6 and 3 months) at the starting point of the intervention, at 3 and 6 months during the dietary intervention with high phenolic EVOO. The correlation of the changes on the lipidemic profile during the survey with the clinical outcome of the patient with CLL was also investigated.
Effect of the dietary intake of high phenolic EVOO on liver function and correlation with the clinical outcome of the patients with CLL | 1 year
  The effect of the dietary intake of high phenolic EVOO on liver function was investigated comparing the biochemical markers of the liver function (Serum glutamic pyruvic transaminase (SGPT (U/L)), Serum glutamic oxaloacetic transaminase (SGOT(U/L) ), lactate dehydrogenase (LDH(U/L)), alkaline phosphatase (ALP(U/L)), gamma-glutamyl transferase (γ-GT(U/L) before the intervention (6 and 3 months) at the starting point of the intervention, at 3 and 6 months during the dietary intervention with high phenolic EVOO. The correlation of the changes on the liver function during the survey with the clinical outcome of the patient with CLL was also investigated.
Effect of the dietary intake of high phenolic EVOO on kidney function and correlation with the clinical outcome of the patients with CLL | 1 year
  The effect of the dietary intake of high phenolic EVOO on kidney function was investigated comparing the conventional biochemical markers of the kidney function Urea(mg/dl) and creatinine (mg/dl ) before the intervention (6 and 3 months) at the starting point of the intervention, at 3 and 6 months during the dietary intervention with high phenolic EVOO. The correlation of the changes on the kidney function during the survey with the clinical outcome of the patient with CLL was also investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Prokopios Magiatis, PhD, Study Director — National and Kapodistrian University of Athens
Locations (1):
- University of Peloponnese, School of Health Sciences, Department of Nursing, Sparti, Lakonias, Greece

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make Individual participant data (IPD) available.

REFERENCES:
- [Background] Parkinson L, Keast R. Oleocanthal, a phenolic derived from virgin olive oil: a review of the beneficial effects on inflammatory disease. Int J Mol Sci. 2014 Jul 11;15(7):12323-34. doi: 10.3390/ijms150712323. PMID 25019344
- [Background] Beauchamp GK, Keast RS, Morel D, Lin J, Pika J, Han Q, Lee CH, Smith AB, Breslin PA. Phytochemistry: ibuprofen-like activity in extra-virgin olive oil. Nature. 2005 Sep 1;437(7055):45-6. doi: 10.1038/437045a. PMID 16136122
- [Background] Pang KL, Chin KY. The Biological Activities of Oleocanthal from a Molecular Perspective. Nutrients. 2018 May 6;10(5):570. doi: 10.3390/nu10050570. PMID 29734791
- [Background] Sabattini E, Bacci F, Sagramoso C, Pileri SA. WHO classification of tumours of haematopoietic and lymphoid tissues in 2008: an overview. Pathologica. 2010 Jun;102(3):83-7. No abstract available. PMID 21171509
- [Background] Hallek M. Chronic lymphocytic leukemia: 2015 Update on diagnosis, risk stratification, and treatment. Am J Hematol. 2015 May;90(5):446-60. doi: 10.1002/ajh.23979. PMID 25908509
- [Background] Rai KR, Sawitsky A, Cronkite EP, Chanana AD, Levy RN, Pasternack BS. Clinical staging of chronic lymphocytic leukemia. Blood. 1975;46(2):219-234. Blood. 2016 Oct 27;128(17):2109. doi: 10.1182/blood-2016-08-737650. No abstract available. PMID 27789434
- [Background] Domen J, Cheshier SH, Weissman IL. The role of apoptosis in the regulation of hematopoietic stem cells: Overexpression of Bcl-2 increases both their number and repopulation potential. J Exp Med. 2000 Jan 17;191(2):253-64. doi: 10.1084/jem.191.2.253. PMID 10637270
- [Background] Marschitz I, Tinhofer I, Hittmair A, Egle A, Kos M, Greil R. Analysis of Bcl-2 protein expression in chronic lymphocytic leukemia. A comparison of three semiquantitation techniques. Am J Clin Pathol. 2000 Feb;113(2):219-29. doi: 10.1309/491W-L1TN-UFQX-T61B. PMID 10664624
- [Background] Wójtowicz, Μ.; Wołowiec, D. Dysregulation of Apoptosis and Proliferation in CLL Cells, in Chronic Lymphocytic Leukemia ed. InTech Rijeka, Croatia. 2012, chapter 3, p37.
- [Background] Gomes LC, Evangelista FCG, Sousa LP, Araujo SSDS, Carvalho MDG, Sabino AP. Prognosis biomarkers evaluation in chronic lymphocytic leukemia. Hematol Oncol Stem Cell Ther. 2017 Jun;10(2):57-62. doi: 10.1016/j.hemonc.2016.12.004. Epub 2017 Feb 1. PMID 28183684
- [Background] Wójtowicz Μ, Wołowiec D (2012). Dysregulation of Apoptosis and Proliferation in CLL Cells, Chronic Lymphocytic Leukemia. www.intechopen.com.
- [Background] Jaiswal PK, Goel A, Mittal RD. Survivin: A molecular biomarker in cancer. Indian J Med Res. 2015 Apr;141(4):389-97. doi: 10.4103/0971-5916.159250. PMID 26112839
- [Background] Peter ME, Hadji A, Murmann AE, Brockway S, Putzbach W, Pattanayak A, Ceppi P. The role of CD95 and CD95 ligand in cancer. Cell Death Differ. 2015 May;22(5):885-6. doi: 10.1038/cdd.2015.25. No abstract available. PMID 25849030
- [Background] Goren L, Zhang G, Kaushik S, Breslin PAS, Du YN, Foster DA. (-)-Oleocanthal and (-)-oleocanthal-rich olive oils induce lysosomal membrane permeabilization in cancer cells. PLoS One. 2019 Aug 14;14(8):e0216024. doi: 10.1371/journal.pone.0216024. eCollection 2019. PMID 31412041
- [Background] Agrawal K, Melliou E, Li X, Pedersen TL, Wang SC, Magiatis P, Newman JW, Holt RR. Oleocanthal-rich extra virgin olive oil demonstrates acute anti-platelet effects in healthy men in a randomized trial. J Funct Foods. 2017 Sep;36:84-93. doi: 10.1016/j.jff.2017.06.046. Epub 2017 Jul 3. PMID 29904393
- [Derived] Rojas Gil AP, Kodonis I, Ioannidis A, Nomikos T, Dimopoulos I, Kosmidis G, Katsa ME, Melliou E, Magiatis P. The Effect of Dietary Intervention With High-Oleocanthal and Oleacein Olive Oil in Patients With Early-Stage Chronic Lymphocytic Leukemia: A Pilot Randomized Trial. Front Oncol. 2022 Jan 21;11:810249. doi: 10.3389/fonc.2021.810249. eCollection 2021. PMID 35127522